CLINICAL TRIAL: NCT07163429
Title: Efficacy of Flurbiprofen Spray for Postoperative Sore Throat Following Double-Lumen Endobronchial Intubation: A Randomized, Double-blind, Controlled Trial
Brief Title: Efficacy of Flurbiprofen Spray for Postoperative Sore Throat Following Double-Lumen Endobronchial Intubation
Acronym: FLURBI-POST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kittitorn Supphapipat, MD (Other)
Responsible Party: Sponsor-Investigator, Kittitorn Supphapipat, MD, Department of Anesthesiology, Faculty of Medicine, Chiang Mai University, Chiang Mai University
Organization: Chiang Mai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ANE-2568-0331
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Post Operative Sore Throat; Hoarseness
Keywords: Postoperative sore throat (POST); Double-lumen intubation; Thoracic surgery; Flurbiprofen spray; Airway complications
MeSH Terms: conditions — Hoarseness | interventions — Flurbiprofen

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either topical flurbiprofen spray or placebo spray applied to the double-lumen tube cuffs before intubation. Outcomes will be assessed at multiple postoperative time points.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flurbiprofen group (Experimental): Participants will receive topical flurbiprofen spray (one spray on the bronchial cuff and two spray on the tracheal cuff, with a total dose of 8.75 mg of flurbiprofen) applied to both the tracheal and bronchial cuffs of the double-lumen tube before intubation
  Interventions: Drug: Flurbiprofen 8.75 MG
- Control group (Placebo Comparator): Participants will receive placebo spray (0.9% normal saline) applied to both the tracheal and bronchial cuffs of the double-lumen tube before intubation.
  Interventions: Drug: Saline spray

INTERVENTIONS:
Drug: Flurbiprofen 8.75 MG — Topical administration of flurbiprofen 8.75 mg spray applied directly to the tracheal and bronchial cuffs of the double-lumen endobronchial tube before intubation. A total of three sprays will be applied: one spray to the bronchial cuff and two sprays to the tracheal cuff, immediately before intubation.
  Other Names: Flurbiprofen spray
  Arms: Flurbiprofen group
Drug: Saline spray — Topical administration of placebo spray (0.9% normal saline) applied in the same manner as the active intervention, with one spray to the bronchial cuff and two sprays to the tracheal cuff of the double-lumen tube before intubation.
  Arms: Control group

SUMMARY:
The goal of this study is to evaluate whether topical flurbiprofen reduces the incidence and severity of postoperative sore throat (POST) and hoarseness in patients undergoing double-lumen tube (DLT) intubation for elective thoracic surgery.

The main question is: Does topical flurbiprofen reduce POST and hoarseness compared with placebo in patients undergoing DLT intubation? Researchers will compare topical flurbiprofen spray with placebo spray.

Participants will:

* Receive a DLT sprayed with either topical flurbiprofen or placebo before intubation.
* Be assessed for POST and hoarseness at 15 minutes, 2 hours, 12 hours, 24 hours, and 48 hours after surgery.

DETAILED DESCRIPTION:
Postoperative sore throat (POST) is a common complication after general anesthesia involving airway manipulation, with reported incidence rates of up to 62%. It includes a spectrum of symptoms such as throat pain, pharyngitis, laryngitis, tracheitis, cough, hoarseness, and dysphagia, typically occurring in the early postoperative period. Although generally self-limiting, severe cases may cause dyspnea and dysphagia, reduce patient satisfaction, and in some cases prolong hospital stay.

POST results from laryngeal and tracheal mucosal injury during tracheal intubation. The pathophysiology is multifactorial, involving direct airway trauma, mucosal irritation and inflammation, ischemia from cuff compression, regurgitation of gastric contents, and gastric tube placement. Risk factors include female sex, younger age, smoking, lung disease, prolonged surgery, patient repositioning, difficult intubation, larger tube diameter, stylet use, high cuff pressure, and frequent suctioning.

The use of double-lumen tubes (DLTs), required for thoracic surgery with one-lung ventilation, has been associated with an even higher incidence of POST due to larger tube size, stylet-assisted insertion, and increased glottic trauma.

Several strategies have been investigated to prevent POST, including cuff pressure control, local anaesthetics, corticosteroids, and nonsteroidal anti-inflammatory drugs (NSAIDs). Dexamethasone and lidocaine have shown some benefit, but results are inconsistent, and POST remains prevalent in clinical practice.

Flurbiprofen, a nonsteroidal anti-inflammatory drug, is available as an oromucosal spray (8.75 mg/dose) and is widely used for sore throat relief in general practice. It reduces airway inflammation and provides analgesia when applied locally. Previous studies suggest that flurbiprofen spray applied to the cuff of laryngeal mask airways or single-lumen tubes reduces POST severity. However, limited evidence is available in the setting of DLT intubation, which carries a higher risk of POST.

This randomized, double-blind, placebo-controlled trial will investigate whether topical flurbiprofen spray applied to the cuff of a DLT before intubation reduces the incidence and severity of POST and hoarseness in patients undergoing elective thoracic surgery. Participants will be randomized to receive either topical flurbiprofen spray or placebo, with outcomes assessed at multiple time points up to 48 hours postoperatively. The study will be conducted at a single academic center, with standardized anesthesia management and blinding of patients, clinicians, and outcome assessors.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 20-80 years
* Undergoing elective thoracic surgery
* Requiring DLT intubation for lung separation
* ASA physical status classification I-III
* Able to communicate and understand the study

Exclusion Criteria:

* Contraindications to use of flurbiprofen, including allergies to flurbiprofen or NSAIDs, active peptic ulcer/ hemorrhage, history of gastrointestinal bleeding or perforation, severe colitis, severe heart failure, chronic kidney disease (CKD) stage IV or end-stage kidney disease (ESRD), or liver failure
* Recent or recurrent upper respiratory tract infection
* History of sore throat or hoarseness within 1 month prior to surgery
* History of previous airway surgery
* Chronic pain conditions
* Pregnancy

Withdrawal criteria

* Fail DLT intubation
* Inability to extubation at the end of surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of POST | Within 48 hours postoperatively
  Presence or absence of postoperative sore throat (POST)

SECONDARY OUTCOMES:
Severity of POST | 15 minutes, 2, 12, 24, and 48 hours postoperatively
  Severity of sore throat measured using a numerical rating scale (0-10) and throat pain scale (TPS: 0 = none, 1 = mild, 2 = moderate, 3 = severe).
Incidence of hoarseness | Within 48 hours postoperatively
  Presence or absence of hoarseness
Severity of hoarseness | 15 minutes, 2, 12, 24, and 48 hours postoperatively
  Severity of hoarseness measured using a 4-point scale (HOAR: 0 = none, 1 = minimal, 2 = moderate, 3 = severe)
Patient satisfaction | 48 hours postoperatively
  Overall patient satisfaction intubation, measured using a 10-point satisfaction scale (0 = not satisfied, 10 = very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Kittitorn Supphapipat, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Chiang Mai University
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Faculty of Medicine, Chiang Mai University, Chiang Mai, Mueang, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared because this is a single-centre investigator-initiated study with a limited sample size, and the data contain potentially sensitive patient information. De-identified summary data may be made available upon reasonable request to the principal investigator

REFERENCES:
- [Background] Uzture N, Menda F, Bilgen S, Keskin O, Temur S, Koner O. The Effect of Flurbiprofen on Postoperative Sore Throat and Hoarseness After LMA-ProSeal Insertion: A Randomised, Clinical Trial. Turk J Anaesthesiol Reanim. 2014 Jun;42(3):123-7. doi: 10.5152/TJAR.2014.35693. Epub 2014 Mar 11. PMID 27366405
- [Background] Mazzotta E, Soghomonyan S, Hu LQ. Postoperative sore throat: prophylaxis and treatment. Front Pharmacol. 2023 Nov 23;14:1284071. doi: 10.3389/fphar.2023.1284071. eCollection 2023. PMID 38074131